CLINICAL TRIAL: NCT03502278
Title: A Lay-Led Intervention for War and Refugee Related Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Seattle Pacific University (Other); Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Lori Zoellner, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 49606; 1R34MH112756 (NIH)
Record Dates: First submitted 2018-03-13; First posted 2018-04-18 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: PTSD
Keywords: refugee
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: A small RCT (N = 60) will be conducted comparing Islamic Trauma Healing in an U.S. Somali refugee sample to a waitlist control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTSD lay-led group treatment program (Active Comparator): This group will go through the Islamic Trauma Healing Program
  Interventions: Behavioral: Islamic Trauma Healing
- Waitlist (No Intervention): Waitlist

INTERVENTIONS:
Behavioral: Islamic Trauma Healing — A lay-led, six-session group intervention that combines empirically supported exposure-based and cognitive restructuring techniques with Islamic principles
  Arms: PTSD lay-led group treatment program

SUMMARY:
This study will examine the initial efficacy and feasibility of a program called Islamic Trauma Healing by conducting a small RCT (N = 60) comparing Islamic Trauma Healing in an U.S. Somali refugee sample to a waitlist control on key targets of PTSD, depression, somatic symptoms, and quality of life. The hypothesis is that those in Islamic Trauma Healing will show a greater reduction of PTSD symptoms, depressive symptoms, and somatic symptoms and show a greater improvement in quality of well-being than those in the waitlist condition (WL).

DETAILED DESCRIPTION:
Islamic Trauma Healing is a lay-led, small-group intervention specifically targeting healing mental wounds of trauma within mosques. The six-session intervention combines empirically supported exposure-based and cognitive restructuring techniques with Islamic principles. A lay-led, group program promotes community building, acknowledges trauma's impact in the community, and facilitates wider implementation. The program is not referred to as "therapy" or "treatment" for "mental illness." It incorporates community building (e.g., shared tea, supplication), integrated Islamic principles that utilize cognitive restructuring through discussion of prophet narratives (e.g., faith during hard times, Prophet Job [Ayyub]), and exposure therapy through individual prayer, talking to Allah about the trauma. Ultimately, the program will follow a self-sustaining train-the-trainer model, led by group leaders, empowering lay leaders to facilitate healing in their communities. Further, training time is dramatically reduced to two, 4-hour training sessions, focusing on teaching skills of group discussion leading rather than training as a lay therapist or mental health counselor. Preliminary data from a community sample and from initial men's and women's groups show a strong perceived need and match with the Islamic faith, with large effects obtained for pre- to post-group across measures (g = 0.76-3.22). Qualitative analysis identified the intervention as operating on potential mechanisms of connectedness to the community, faith integration, healing, and growth. The preliminary data point to the program being well-received and offering a promising model for delivery of a trauma-focused intervention to Muslim communities. The next steps are examining Islamic Trauma Healing in a RCT, further isolating mechanisms of change, and ascertaining feasibility for wider dissemination studies.

ELIGIBILITY:
Inclusion Criteria:

* Experienced a DSM-5 trauma at least 12 weeks ago
* Report current re-experiencing or avoidance symptoms
* Somali background
* Islamic faith
* 18-65 year of age

Exclusion Criteria:

* Immediate suicide risk, with intent or plan
* Cannot understand consent/visible cognitive impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2018-07-14 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
PTSD Scale - Self-Report for DSM-5 (PS-SR-5; Foa et al., 2015 | 3 Month Follow-up
  PTSD symptoms will be measured using the PTSD Scale - Self-Report for DSM-5 (PS-SR-5; Foa et al., 2015). Twenty items comprise the PTSD severity scale, with scores ranging from 0 to 80 and higher scores indicating higher PTSD severity. A total score is calculated.

SECONDARY OUTCOMES:
Depression symptoms will be measured using the Patient Health Questionnaire-9 (PHQ-9; Kroenke, Spitzer, & Williams, 2001) | 3 Month Follow-up
  The PHQ-9 is a self-report measure of depression symptoms with each question rated from 0-3.
Somatic symptoms will be measured using the Patient Health Questionnaire-15 (PHQ-15; Kroenke, Spitzer, & Williams, 2002) | 3 Month Follow-up
  The PHQ-15 is a self-report assessment of somatic symptoms (e.g., stomach pain, headaches, dizziness) .
Quality of well-being Index | 3 Month Follow-up
  The WHO-5 Wellbeing Index (WHO-5; Bech, Olsen, Kjoller, & Rasmussen, 2003) will be used to measure well-being. This five-item measure assesses emotional well-being on a 0-5 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lori A Zoellner, PhD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Case Western Reserve University, Cleveland, Ohio
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with the NIMH Data Archive
Supporting Information: Study Protocol, SAP
Time Frame: Per requirements of the NIMH Archive.
Access Criteria: Per requirements of the NIMH Archive.

REFERENCES:
- [Derived] Zoellner LA, Bentley JA, Musa K, Mohamed F, Ahmed LB, King KM, Feeny NC; Islamic Trauma Healing Clinical Team. Lay-Led Intervention for War and Refugee Trauma: A Randomized Clinical Trial. JAMA Netw Open. 2024 Aug 1;7(8):e2429661. doi: 10.1001/jamanetworkopen.2024.29661. PMID 39186273

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT03502278/Prot_SAP_002.pdf